CLINICAL TRIAL: NCT05435274
Title: A Phase 1/2, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of HS-10376 Monotherapy in Patients With Advanced Non-small-Cell Lung Cancer
Brief Title: Phase 1/2 Study of HS-10376 in Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-10376-101
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Advanced Non-Small-Cell Lung Cancer
Keywords: NSCLC; Non-Small Cell Lung Cancer; HS-10376; EGFR/HER2 Exon 20 insertion mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10376 (Experimental): Phase 1a：Dose Escalation：Subjects with advanced NSCLC will be enrolled in dose escalation cohorts. Dose escalation of HS-10376 will be done to determine maximum tolerated dose.
  Phase 1b：Dose Expansion：Depending on data obtained from the dose escalation part, dose expansion may proceed with multiple cohorts in subjects with advanced NSCLC having a EGFR/HER2 Exon 20 insertion mutation.
  Phase 2：Subjects with locally advanced or metastatic EGFR Exon 20 insertion NSCLC will be enrolled in phase 2 part to evaluate the efficacy and sufficient safety of HS-10376 as monotherapy.
  Interventions: Drug: HS-10376

INTERVENTIONS:
Drug: HS-10376 — HS-10376 will be administered orally once daily in a continuous regimen

SUMMARY:
HS-10376 is an oral, highly selective, small molecular inhibitor of EGFR/HER2 Exon 20 insertion mutation. This study will evaluate the safety, tolerability, pharmacokinetics and clinical activity of HS-10376 in Chinese advanced Non-Small Cell Lung Cancer (NSCLC) patients.

DETAILED DESCRIPTION:
This is a phase 1/2, first-in-human, open-label, multicenter study of HS-10376, this study has two parts: phase 1 and phase 2. The phase 1 portion consists of dose escalation and dose expansion, which is aimed to assess the safety and tolerability of HS-10376 in subjects with advanced NSCLC and evaluate the preliminary efficacy of HS-10376. Phase 2 will be conducted to evaluate the efficacy of HS-10376 in subjects with locally advanced or metastatic NSCLC with a EGFR Exon 20 insertion mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women greater than or equal to 18 years
2. Locally advanced or metastatic NSCLC patients confirmed by histology or cytology, for which standard treatment is invalid, unavailable or intolerable
3. Pathological, tumor tissue samples can be used to test EGFR/HER2 Exon 20 insertion mutation by central laboratory for subjects
4. At least one measurable lesion in accordance with RECIST 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0~1
6. Estimated life expectancy >12 weeks
7. Reproductive-age women agree to use adequate contraception and cannot breastfeed while participating in this study and for a period of 6 months after the last dose. Likewise, men also consent to use adequate contraceptive method within the same time limit.
8. Females must have the evidence of non-childbearing potential
9. Signed and dated Informed Consent Form

Exclusion Criteria:

1. Treatment with any of the following:

   * Previous or current treatment with EGFR Exon 20 insertion inhibitors, HER2 Exon 20 insertion inhibitors or EGFR/HER2 Exon 20 insertion inhibitors
   * Any cytotoxic chemotherapy, anticancer Chinese medicine and targeted small molecule inhibitors within 14 days of the first dose of HS-10376
   * Any investigational agents and large molecule antibodies within 28 days of the first dose of HS-10376
   * Local radiotherapy for palliation within 2 weeks of the first dose of HS-10376, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks of the first dose of HS-10376
   * Major surgery (including craniotomy, thoracotomy, or laparotomy, etc.) within 4 weeks of the first dose of HS-10376
2. Inadequate bone marrow reserve or serious organ dysfunction
3. Uncontrolled pleural, ascites or pericardial effusion
4. Untreated, symptomatic or active central nervous system metastases
5. Severe or poorly controlled hypertension
6. Immunodeficiency disease and active infectious disease
7. Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow oral medications
8. History of hypersensitivity to any active or inactive ingredient of HS-10376 or to drugs with a similar chemical structure or drugs belonging to the same category of HS-10376
9. The subject who is unlikely to comply with study procedures, restrictions, or requirements judged by the investigator
10. The subject whose safety cannot be ensured or study assessments would be interfered judged by the investigator
11. Pregnant women, breastfeeding women or woman who has a child-bearing plan during the study
12. History of neuropathy or mental disorders, including epilepsy and dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-10-07 (Estimated); Study Completion 2025-10-07 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD)-Part Ia | From the single dose to the last dose of the first cycle defined as 21 days of multiple dosing (total 28 days)
  Number of participants with dose limiting toxicity
To evaluate clinical activity/efficacy of HS-10376 by assessment of objective response rate-Phase Ib/II | up to 24 months
  Objective response rate (ORR) assessed by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Number of participants with treatment related adverse events | From baseline until 28 days after the last dose
  Number of participants with treatment related adverse events.
Observed maximum plasma concentration (Cmax) after single dose of HS-10376 | From pre-dose to 120 hours after single dose on Day 1
  In the study of single-dose, Cmax will be obtained following administration of a single oral dose of HS-10376
Time to reach maximum plasma concentration (Tmax) after single dose of HS-10376 | From pre-dose to 120 hours after single dose on Day 1
  In the study of single-dose, Tmax will be obtained following administration of a single oral dose of HS-10376
Apparent terminal half-life (T1/2) after single dose of HS-10376 | From pre-dose to 120 hours after single dose on Day 1
  Apparent terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Duration of response (DOR) | 24 months
  DOR assessed by RECIST 1.1 criteria
Disease Control Rate (DCR) | 24 months
  DCR assessed by RECIST 1.1 criteria
Progression-free survival (PFS) | 24 months
  PFS assessed by RECIST 1.1 criteria
Overall survival (OS) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No